CLINICAL TRIAL: NCT01308229
Title: Assessment of the Safety and Efficacy of the Nile PAX® Drug Eluting Coronary Bifurcation Stent System for the Treatment of Single de Novo Bifurcation Lesions in Native Coronary Arteries
Brief Title: Safety and Efficacy Study of the Nile PAX Drug-Eluting Coronary Bifurcation Stent
Acronym: BIPAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MINVASYS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIN0803
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Disease
Keywords: Bifurcation; Dedicated; Drug-eluting stent; Angioplasty; Coronary artery disease; Coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nile PAX® (Experimental)
  Interventions: Device: Nile PAX® paclitaxel-eluting coronary stent

INTERVENTIONS:
Device: Nile PAX® paclitaxel-eluting coronary stent — Implantation of a Nile PAX bifurcation dedicated drug-eluting stent in coronary arteries to treat stenosis lesions

SUMMARY:
The purpose of this trial is to assess the safety and efficacy of the Nile PAX® Drug Eluting Coronary Bifurcation Stent System for the treatment of single de novo bifurcation lesions in native coronary arteries with a main branch reference vessel diameter of 2.5-3.5 mm and side branch reference vessel diameter of 2.0-3.0 mm.

DETAILED DESCRIPTION:
The BIPAX clinical trial is a prospective, non-randomized, multicenter, clinical trial evaluating the investigational coronary bifurcation device Nile PAX® in patients with main branch reference vessel diameters >= 2.5 mm and <= 3.5 mm, side branch reference vessel diameters >= 2.0 and <= 3.0 and lesion length <= 14 mm. The trial allows the treatment of a single de novo bifurcation lesion in native coronary arteries following the provisional T-stenting technique with mandatory pre-dilatation of the main branch. In case the side branch requires a stent the treatment will be completed when possible with a Delta PAX® Drug Eluting Side Branch Stent.

The BIPAX clinical trial will enroll 100 patients. All patients will receive Quantitative Coronary Angiography (QCA) after stent implantation and at 9 months follow-up. All patients will have a clinical follow-up at 1, 6, 9 and 12 months and subsequently every year up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* De novo bifurcation lesions following the Medina classification except (0,0,1).
* Maximum one bifurcation lesion per patient.
* Single bifurcation lesion per vessel.
* The patient is at least 18 years of age. The patient has clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, or a positive functional trial.
* The patient is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergent coronary artery bypass graft (CABG) surgery.
* The patient or patient's legal representative has been informed of the nature of the trial and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical site.
* The patient agrees to return to the same research facility for all required post-procedure follow-up visits.

Exclusion Criteria:

* De novo bifurcation lesion Medina (0,0,1).
* Left main bifurcation.
* Heavily calcified lesions.
* Severe tortuous lesions.
* Documented left ventricular ejection fraction (LVEF) < 30% at most recent evaluation.
* Women of childbearing potential.
* Chronic total occlusion (CTO).
* Previous PCI of the target lesion.
* Second lesion requiring treatment in target vessel.
* Second bifurcation lesion requiring treatment.
* Currently participating in an investigational drug or another device trial that has not completed the primary endpoint or that clinically interferes with the current trial endpoints; or requires coronary angiography, IVUS or other coronary artery imaging procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Angiographic restenosis rate (%) | 9 months post-procedure
  Angiographic restenosis rate of the main branch and side branch by Quantitative Coronary Angiography (QCA).

SECONDARY OUTCOMES:
Clinically-driven Target Vessel Failure (TVF) | 9 months post-procedure
Target Lesion Revascularization (TLR) | 9 months after procedure
Target Vessel Revascularization (TVR) | 9 months post-procedure
Acute success (device, lesion, and procedure) | at procedure
Angiographic in-stent Late Lumen Loss (LLL) | 9 months post-procedure
Minimum luminal diameter (MLD) | 9 months post-procedure
Angiographic parameters | 9 months post-procedure
  Angiographic parameters (in-stent and in-segment) including percent Diameter Stenosis (%DS)
Major Adverse Cardiac Event (MACE) rate | 30 days and 9 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jean FAJADET, MD, Principal Investigator — Clinique Pasteur Toulouse
Locations (10):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Tokuda Hospital, Sofia, Bulgaria
- France (4):
  - Centre Cardiologique d'Evecquemont, Évecquemont
  - Clinique Saint Hilaire, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Pasteur, Toulouse
- Casa di Cura Montevergine, Mercogliano, Italy
- Thorax Centre, Rotterdam, Netherlands
- Karol Marcinkowski University of Medical Sciences, Poznan, Poland
- Hospital Universitari Vall D´Hebron, Barcelona, Spain